CLINICAL TRIAL: NCT07232186
Title: The Effect of the NURSIM-KID (NURSE IMAGE-KID) Program for Hospitalized Migrant Children on the Nursing Image of Children and Parents: A Randomized Controlled Trial
Brief Title: The Effect of the NURSIM-KID Program for Migrant Children Hospitalized in Hospitals on the Nursing Image of Children and Parents
Acronym: NURSIM-KID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Bahar Aksoy, PhD, Akdeniz University Kumluca Health Science Faculty
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Akdeniz Üniversitesi
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hospitalized Migrant Child; Migrant Parent and Child
Keywords: Child, Hospitalized; Child, Migrant; Nursing Care; Nurse-Patient Relations; Professional Image; Parental Attitudes; Program Evaluation

STUDY DESIGN:
Intervention Model Description: This study is a parallel group randomized controlled trial.Children and their mothers who meet the inclusion criteria at the pediatric ward at the time of the study will be interviewed. Prior to randomization, they will be informed about the study and their consent will be obtained, and data on the children's characteristics will be collected. The intervention group of the study consists of children and families who will receive NURSIM-KID training, while the control group consists of children and families who are informed in accordance with clinical routine. To prevent selection and detection bias in the study, participants will be randomly assigned to the intervention and control groups by a statistician outside of the research team. The "block randomization" method, one of the "fixed probability randomization" methods, will be used for randomization in this study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NURSIM-KID Program (Experimental): Participants assigned to the experimental group will receive the NURSIM-KID (Nursing Image for Kids) program in addition to routine hospital care. Participants will be assigned to this group through randomization.
  Interventions: Behavioral: NURSIM-KID Program
- Routine Hospital Care (No Intervention): Participants in the control group will receive routine hospital care only, with no additional educational or behavioral intervention. Routine care includes standard nursing care provided by the hospital team. Participants will be assigned to this group through randomization.

INTERVENTIONS:
Behavioral: NURSIM-KID Program — The NURSIM-KID program is a three-day structured intervention designed to support 8-11-year-old hospitalized children's perceptions of the nursing profession. It introduces children to the hospital environment, the nurse's role, and common medical equipment in a simple, child-friendly manner. Through puppets and the picture book "Who Am I? Nurse," children learn about nursing care, empathy, and communication. The program emphasizes emotional safety and active participation, encouraging children to express their feelings and questions. On the final day, children receive a participation certificate, reinforcing positive and trusting attitudes toward nurses and healthcare.
  Arms: NURSIM-KID Program

SUMMARY:
The nursing profession has a dynamic image in society, shaped by individuals' lives, cultural backgrounds, and interactions with healthcare services. The image of nursing formed during childhood, in particular, directly influences individuals' attitudes toward healthcare professionals and their participation in healthcare services. Migrant children, however, may perceive the nursing profession in a more limited and negative context due to reasons such as unfamiliarity with the hospital environment, language barriers, and cultural differences. Based on this, the aim of this study is to evaluate the effect of the NURSIM-KID program, developed for migrant children aged 8-11 years receiving inpatient treatment in the pediatric ward of Kilis Prof. Dr. Alaeddin Yavaşca State Hospital, on the images of the nursing profession held by children and their parents. The program aims to contribute to introducing the nursing profession in a more positive and functional way, using methods appropriate to the children's age and developmental level. The limited number of studies in the literature addressing the perceptions of migrant children and their parents regarding the image of nursing highlights the importance of this research and the original contribution it will make to the field. The findings of the study are of a nature that could guide the development of nursing education, child-friendly hospital practices, and culturally supportive initiatives.

DETAILED DESCRIPTION:
Migrant children often experience illness and hospitalization more traumatically than their peers due to socioeconomic difficulties, language barriers, cultural adaptation problems, and limited access to health services. Hospitalization can trigger loneliness, insecurity, and fear, while language barriers hinder self-expression and communication with healthcare staff. Cultural differences may make the hospital environment and medical procedures appear confusing or threatening, and parents' limited participation in care can deprive children of emotional support. Top (2023) identified language barriers, cultural differences, hygiene practices, low health literacy, and poor post-discharge care continuity as major challenges in caring for hospitalized migrant children. These factors complicate both children's treatment and nursing care delivery. The first interaction between migrant children and nurses plays a key role in shaping their image of the nursing profession. Nursing image is a dynamic, multidimensional concept that changes over time depending on one's social environment, culture, and experiences. According to Boulding's (1956) image theory, people's perceptions of a profession are shaped by their experiences and the messages they receive about it. Children, therefore, form their perceptions of nursing through direct hospital experiences, serving as neutral reflectors of professional image. However, existing studies have mostly focused on children's hospital experiences or satisfaction with nursing care, with limited research exploring their lasting impressions of the profession. For migrant children, the image of nursing is particularly affected by communication difficulties, cultural differences, and healthcare providers' attitudes. In a study by Güney, Düzkaya, and Uysal (2025), nurses reported challenges such as miscommunication, culturally inappropriate practices, patient safety concerns, time loss, and emotional fatigue while caring for migrant children. These challenges can lead children to perceive nursing as a distant, procedure-oriented profession that lacks communication and empathy. Negative perceptions, in turn, may reduce children's willingness to cooperate and engage in care. Yet, the image of nursing formed in childhood can significantly influence individuals' later attitudes toward healthcare services, their health literacy, and even career choices. Based on the ecological systems theory, individuals' behaviors are shaped by their broader social and familial contexts. Similarly, control systems theory emphasizes the importance of parent-child interactions in shaping attitudes and behaviors. Therefore, parents' perceptions of nursing indirectly influence their children's image of the profession. A multicenter study conducted in Türkiye found that children generally held more positive images of nursing than their parents, but parental attitudes remained an important determinant of these perceptions. Given these dynamics, structured programs that provide positive and meaningful encounters with nursing during hospitalization are essential for migrant children. The NURSIM-KID (Nursing Image for Kids) program was designed to assess and improve the nursing image among hospitalized migrant children aged 8-11 years. By introducing nursing in an interactive, age-appropriate, and culturally sensitive manner, the program aims to portray nurses as caregivers who provide support, trust, and compassion-not merely as medical professionals. Ultimately, NURSIM-KID seeks to identify negative perceptions early and foster positive, lasting attitudes toward nursing and healthcare among migrant children.

ELIGIBILITY:
Inclusion Criteria:

The child must be between the ages of 8 and 11. The child must be hospitalized for at least 3 days. The child must not have any auditory, visual, speech, or mental disabilities. Both the parent and the child must volunteer to participate in the study. Parents and children who can read Turkish and have communication skills will be included in the study.

Exclusion Criteria:

Parents who do not agree to participate in the study. Parents and children who do not have communication skills in Turkish will not be included in the study.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Child-Parent Introductory Information Form | Before starting the study
  This form was designed to collect basic information about the demographic characteristics and hospital experiences of the participating children and their parents. Developed by the researchers in line with relevant literature (Cırık et al., 2024; Cırık et al., 2025), the form consists of both closed-ended and open-ended questions. The form assesses the children's sociodemographic characteristics, such as age, gender, and educational status, as well as their past health-related experiences. It also includes questions about the child's current health status, previous hospitalizations, and experiences related to the hospital environment. The section for parents includes closed-ended questions to assess their age, educational status, employment status, family structure, health status, and perceptions and attitudes toward the nursing profession

SECONDARY OUTCOMES:
Nursing Image Perceived by Children Scale | At study initiation, the researcher administers the Children's Perceived Nursing Image Scale as a pre-test; the same scales are reapplied on Day 3 to collect post-test data
  The "Nursing Image Perceived by Children Scale" used in this study was developed by Apaydın Çirik et al. (2025) to assess the perceptions of children aged 8-11 years regarding the nursing profession. The scale consists of 35 items and is administered using a 5-point Likert-type rating system. Participants score each statement from "strongly disagree" to "strongly agree." There are no reverse-scored items. The scale consists of four subscales: professional duties and responsibilities, professional image, perception, and communication. Possible scores range from 35 to 175, with higher scores indicating a more positive image of the nursing profession. As a result of the validity and reliability analyses conducted in the development study, the scale was accepted as a valid and reliable measurement tool for children aged 8-11 years in Turkish society. The total Cronbach alpha coefficient of the scale was calculated as 0.93.
Nursing Image Scale | At study initiation, the researcher administers the Nursing Image Scale and the Children's Perceived Nursing Image Scale as a pre-test; the same scales are reapplied on Day 3 to collect post-test data
  This scale was developed to assess individuals' perceptions of the nursing profession. The Nursing Image Scale (NUS) was developed by Özsoy (2000) and adapted into Turkish by Çınar and Demir (2009). The scale consists of 28 items and three subscales: overview (7 items), communication (6 items), and professional-educational competencies (15 items). Items are answered on a three-point Likert-type scale: "1 = Disagree," "2 = Partly Agree," and "3 = Agree." Some items are reverse-scored. The total score ranges from 28 to 84, with higher scores reflecting a more positive image of the nursing profession. The Cronbach alpha internal consistency coefficient of the scale was reported as 0.70 in the original study. In the Turkish adaptation study, the alpha values for the sub-dimensions ranged from 0.60 to 0.75, and the test-retest reliability was 0.70.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guney A, Sonmez Duzkaya D, Uysal G. Pediatric Nurses' Experiences in Refugee Children Care: A Qualitative Research. Disaster Med Public Health Prep. 2025 Apr 15;19:e96. doi: 10.1017/dmp.2025.87. PMID 40230245
- [Result] Uzun LN. The effect of creative drama on nursing image: Randomized controlled study. Nurse Educ Pract. 2024 May;77:103970. doi: 10.1016/j.nepr.2024.103970. Epub 2024 Apr 17. PMID 38678868
- [Result] Ustuner Top F. The Challenges in the Care of Immigrant Children in the Clinic: A Phenomenological Study. J Pediatr Health Care. 2023 Sep-Oct;37(5):492-500. doi: 10.1016/j.pedhc.2023.03.005. Epub 2023 Apr 7. PMID 37031099
- [Result] Cirik VA, Aksoy B, Gul U. The image of nursing in the eyes of Generation Alpha and their parents in Turkiye: A multicenter cross-sectional survey. J Pediatr Nurs. 2024 Sep-Oct;78:124-132. doi: 10.1016/j.pedn.2024.06.018. Epub 2024 Jun 24. PMID 38917614
- [Result] Apaydin Cirik V, Aksoy B, Bektas M. Development of Children's Perceived Nursing Image Scale: A Validity and Reliability Study. J Eval Clin Pract. 2025 Feb;31(1):e14315. doi: 10.1111/jep.14315. PMID 39831646